CLINICAL TRIAL: NCT06476951
Title: The Effects of Parent-Child Activity Program on Physical Activity of Children With Cancer
Brief Title: The Effects of Parent-Child Activity Program on PA of Children With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ke Liu (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Ke Liu, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: L2023SYSU-HL-020; SYSKY-2024-148-02 (Registry Identifier: SYSKY-2024-148-02)
Record Dates: First submitted 2024-06-11; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Childhood Cancer; Physical Activity; Intervention Program; Parent-Child Relations
Keywords: Childhood Cancer; Physical Activity; Parent-Child Activity Program
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): No specific care in physical activity
- Parent-Child Physical Activity Program (Experimental): Parent-Child Physical Activity Program
  Interventions: Behavioral: Parent-Child Physical Activity Program

INTERVENTIONS:
Behavioral: Parent-Child Physical Activity Program — The program includes online education, parent-child games, parent-child dancing, and other parent-child physical activity activities.
  Arms: Parent-Child Physical Activity Program

SUMMARY:
The goal of this clinical trial is to test the effect of Parent-Child activity program on physical activity of children with cancer. The main question it aims to answer is:

* Whether the Parent-Child activity program has effectiveness for children with cancer on their physical Activity, Physical Activity Self-Efficacy, Physical Activity Enjoyment, Family Support, and for parents on Physical Activity based on the Youth Physical Activity Promotion Model.

Participants will:

* Receive a handbook on information related to physical activity and Parent-Child physical activity when the child is undergoing treatment.
* Participate in Parent-Child activities, such as throw ball catch game, which are organized by the professionals.
* Parents or/and children receive subscriptions on physical activity through WeChat, including the benefits of physical activities and Parent-Child activities, common physical activities and Parent-Child activities, and follow-up video.

Researchers will compare control group to see if there are differences between usual care on physical activity and Parent-Child activity program

DETAILED DESCRIPTION:
The intervention includes three main contents:

1. Establishment and use of WeChat group - information support Nurses in the intervention group establish a WeChat group and invite children with cancer and/or their parents to join the WeChat group, and the children and their parents were regularly subscribed the knowledge related to physical activity on a weekly basis. The contents mainly include the following modules: ① the benefits and importance of physical activity for patients with cancer and the harm of sedentary activities; ② the expert advice and guidelines on physical activity for patients with cancer; ③ common types of physical activities for children with cancer; ④ the suitable amount, frequency and intensity of physical activities for children with cancer; ⑤ the important role of the parents in their children's physical activities and the significance of parent-child activities; ⑥ the measures to ensure the safety of the children during the course of their physical activities; ⑦ emergency treatment plan for any uncomfortable symptoms. In addition, every Monday morning at 8 a.m., the researcher sent a physical activity record list to them, inviting children and parents to record the physical activity accordingly, in order to calculate the amount of exercise per week.
2. Use of WeChat Official account - information and skills support Using the WeChat Official account of the hospital's Department of Paediatric Oncology, tweets and video content related to physical activity are published every Thursday, Saturday and Sunday, mainly including knowledge of physical activity and videos on common types of physical activity and parent-child physical activity. Demonstrations and follow-up exercises videos are provided so that children and parents can choose suitable physical activities for exercise according to their own physical conditions and preferences. Among them, the knowledge of the benefits of physical activity, the importance and significance of parent-child activities and how to ensure safety during exercise; physical activity videos include: ① common warm-up and stretching exercises and action points; ② common aerobic exercises (such as brisk walking, jogging, cycling, jumping rope, aerobics, etc.) and action points; ③ common resistance exercises (such as sit-ups, push-ups, high leg lifts, dumbbell exercises, etc.) and action points; ③ common resistance exercises (such as sit-ups, push-ups, high leg lifts, dumbbell exercises, etc.) and action points. (e.g. sit-ups, push-ups, elevated leg exercises, dumbbell exercises, etc.) and the main points of the movements; (4) common parent-child activities (e.g. relay running, two-person aerobics, two-person games, ball games, swinging sports, jumping grids, throwing sandbags, jumping hoops, etc.) and the main points of the movements; (5) common outdoor family sports (e.g. mountain climbing, rowing, etc.) and the strategies and precautions.
3. Face-to-face parent-child group activities - venue support The children and their parents were told to follow up for every 4 weeks, and on the day of their return to the hospital for review, 5-7 pairs of children and their parents from the review were organised to participate in face-to-face parent-child group activities together for 90-120 minutes each time. The researcher provided them with venues and sports items (e.g., jump ropes, batons, elastic bands, sports videos, etc.), and organised them to participate in parent-child activities and competitions by using open, flat and safe venues in the hospital. The main contents of the group parent-child activities included: ① warm-up and stretching activities (following the demonstration exercises); ② parent-child games and competitions: such as jumping lattice, relay running, wooden man, throwing sandbags, badminton, ball-carrying running, tug-of-war, etc.; and③parent-child dance demonstration and evaluation.

The intervention will last for 12 weeks, and followed up will be organized for 3 months after the completion of all interventions.

ELIGIBILITY:
Inclusion Criteria of children:

* aged 6-14 years when they are recruited
* diagnosed with cancer
* are undergoing cancer treatment when they are recruited
* are able to communicate in Chinese

Exclusion Criteria of children:

* have physical impairment
* have cognitive impairment
* have impaired mental status

Inclusion Criteria of parents:

* are able to communicate in Chinese and read Chinese
* are able to use a smart phone with the instant messaging application WeChat

Exclusion Criteria of parents:

* have emotional or psychiatric disorders
* have cognitive problems

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Children's Leisure Activities Study Survey Chinese | At baseline, and 1, 2, 3 months during the intervention, and 3 months after intervention
  To calculate the time that children spend in sedentary behavior, low-intensity physical activity, and moderate-to-vigorous physical activity in last seven days.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | At baseline, and 1, 2, 3 months during the intervention, and 3 months after intervention
  To calculate the time that parents spend in sedentary behavior, low-intensity physical activity, and moderate-to-vigorous physical activity in last seven days.
Shortened Chinese Version Physical Activity Self-efficacy Scale | At baseline, and 1, 2, 3 months during the intervention, and 3 months after intervention
  To measure the physical activity self-efficacy of children with cancer. Higher scores mean a better outcome.
Short-form Physical Activity Enjoyment Scale | At baseline, and 1, 2, 3 months during the intervention, and 3 months after intervention
  To measure the enjoyment of physical activity in children with cancer. Higher scores mean a worse outcome.
the Social Support for Physical Activity Scale | At baseline, 3 months during the intervention, and 3 months after intervention
  To measure the perceived family support of physical activity in children with cancer. Higher scores mean a better outcome.
Body mass index (BMI) | At baseline, 3 months during the intervention, and 3 months after intervention
  Weight in kilograms, height in meters and weight and height will be combined to report BMI in kg/m^2
Body fat mass | At baseline, 3 months during the intervention, and 3 months after intervention
  Weight of body fat mass in kilograms
Muscle | At baseline, 3 months during the intervention, and 3 months after intervention
  Weight of muscle mass in kilograms
Body fat percentage | At baseline, 3 months during the intervention, and 3 months after intervention
  Body fat percentage in percentage
Muscle percentage | At baseline, 3 months during the intervention, and 3 months after intervention
  Muscle percentage in percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT06476951/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT06476951/ICF_001.pdf